CLINICAL TRIAL: NCT05639738
Title: An Exploratory and Monocentric Study to Assess Clinical, Biological and Biometrological Paramaters in Adult Subjects With Mild to Moderate Atopic Dermatitis (AD)
Brief Title: Assessment of Clinical, Biological and Biometrological Paramaters in Adult Subjects Suffering From AD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADFLAREPREDICT
Record Dates: First submitted 2022-09-16; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subject (Other): Clinical and instrumental measurements
  Interventions: Other: Clinical and instrumental measurements

INTERVENTIONS:
Other: Clinical and instrumental measurements — * Clinical evaluations
  * Non-invasive instrumental measurements
  * Subject's evaluations

SUMMARY:
The aim of the study is to collect different parameters (clinical, biological and biometrological) of Atopic Dermatitis (AD) in order to identify which factors are modified during the flare-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged between 18 to 50 years included
* Subject suffering from Atopic Dermatitis according to the "U.K. Working Party's Diagnostic Criteria for Atopic Dermatitis" (6)
* Subject with mild to moderate Atopic Dermatitis with 20 <= SCORAD <= 40 at inclusion
* Subject with flare frequency ≥ 4 on the target areas over the last year
* Subject with a cutaneous target area, allowing the measurements, located on upper or lower limbs and defined as a usual AD flare area according to the subject
* Subject with a target area with 22 <= target SCORAD signs <= 10 following:

  * Erythema ≥ 1
  * Dryness ≥ 1 1
* Subject with a control area, allowing the measurements, located on upper or lower limbs and defined as :

  * A non- usual AD flare area according to the subject and the investigator
  * A sufficient distance from the cutaneous target area according to the investigator

Exclusion Criteria:

* Subject with a surinfected AD
* Subject having any other dermatologic condition other than AD or characteristics (e.g: tatoo) on the target area liable to interfere with the study assessments
* Subject with another dermatologic condition, acute or chronic or disease or history of disease considered by the investigator, liable to interfere with the study assessments, or hazardous for the subject or incompatible with the study according to the investigator
* Any surgical intervention on upper or lower limbs during the previous weeks or months liable to interfere with the study data according to the investigator
* Systemic immunosuppressive therapy (excepted systemic corticoids) within 3 months before the inclusion visit or ongoing at inclusion visit (except during flare period)
* Systemic corticoids taken within 4 weeks before the inclusion visit or ongoing at inclusion visit (except during flare period)
* Phototherapy performed within 4 weeks before the inclusion visit or ongoing at inclusion visit (except during flare period)
* Systemic antibiotics taken within 7 days before the inclusion visit or ongoing at inclusion visit (except during flare period)
* Moderate to high-potency topical corticosteroids applied within 7 days on upper or lower limbs before the inclusion visit or ongoing at inclusion visit (except during flare period)
* Topical immunomodulators, applied within 7 days on upper or lower limbs before the inclusion visit or ongoing at inclusion visit (except during flare period)
* Topical or oral treatment instaurated or modified before the inclusion visit or planned to be instaurated during the study or ongoing at inclusion visit, liable to interfere with the study, according to the investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Assessment of clinical parameters in Atopic Dermatitis during and outside flares-up | Change from baseline to 3 months
  * SCORAD (SCOring Atopic Dermatitis) and PO-SCORAD (Patient Oriented SCORing Atopic Dermatitis) are a scoring system based on the assessment of extent and intensity in a standardized manner
  * Target SCORAD is the sum of all SCORAD objective signs scores: erythema, oedema/papulation, oozing/crusts, excoriation, lichenification and dryness evaluated on a target area
Colonization of microorganisms involved in Atopic Dermatitis flares-up from PCR analysis on a swab sample | Change from baseline to 3 months
  Colonization of microorganisms will be expressed by percentage of each microorganism
Assessment of lipids profiles in Atopic Dermatitis by mass spectroscopy from swab samples | Change from baseline to 3 months
  Each characteristic peak corresponding to specific lipid will be quantified by its mass intensity
Assessment of cutaneous hydratation in Atopic Dermatitis during and outside flares-up | Change from baseline to 3 months
  Cutaneous hydration evaluated by humidity of the stratum corneum. The measurement is based on capacitance measurement of the stratum corneum.
Assessment of skin barrier condition in Atopic Dermatitis during and outside flares-up | Change from baseline to 3 months
  The measurement is based on Trans-Epidermal Water Loss measurement
Assessment of pH in Atopic Dermatitis during and outside flares-up | Change from baseline to 3 months
  pH evaluated by a pH-meters
Assessment of erythema in Atopic Dermatitis during and outside flares-up | Change from baseline to 3 months
  Assessment the color of the surface of the skin

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche sur la Peau, Toulouse, France